CLINICAL TRIAL: NCT00452621
Title: A Phase IV, Uncontrolled, Open-Label, Multi-Center Study in Children and Adolescents: Evaluation of Long-Term Immunogenicity in Subjects Boosted With a New Pediatric TBE Vaccine (Free of Protein-Derived Stabilizer) in Study V48P4E1, Five Years After First Booster Immunization
Brief Title: Evaluation of Long-Term Immunogenicity in Children and Adolescents Boosted With a New Pediatric TBE Vaccine After Five Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V48P4E3
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-04

CONDITIONS: Encephalitis, Tick-Borne
Keywords: blood draw five years after booster-immunization with TBE vaccine to investigate immunogenicity in children; TBE
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — Blood Specimen Collection

INTERVENTIONS:
Procedure: blood draw

SUMMARY:
blood draw five years after booster-immunization with TBE vaccine to investigate immunogenicity in children

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes aged >1 years at the time of enrollment in V48P4 who participated in studies V48P4E1 and V48P4E2, and who/whose parents or legal guardians are willing to sign informed consent.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 235 (Estimated)
Dates: Start 2007-02

PRIMARY OUTCOMES:
1) To investigate the kinetics of the immune response of subjects who participated in studies V48P4 (primary immunization), V48P4E1 (first booster immunization) and V48P4E2 (serological follow-up) with respect to antibody titers in terms of:· percentage

SECONDARY OUTCOMES:
(2) To investigate the kinetics of the immune response of subjects who participated in studies V48P4 (primary immunization), V48P4E1 (first booster immunization) and V48P4E2 (serological follow-up) in terms of:· percentage of subjects with antibody conce

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis
Locations (8):
- Germany (8):
  - Center 7, Aschaffenburg
  - Center 2, Bobingen
  - Center 11, Eberbach /Neckar
  - Center 4, Kaufering
  - Center 15, Pegnitz
  - Center 1, Weilheim I. OB
  - Center 8, Wiesloch
  - Center 16, Zirndorf